CLINICAL TRIAL: NCT00549003
Title: Efficacy and Cost Effectiveness of Malaria Diagnosis Procedures and the Rational Use of ACT in Zanzibar
Acronym: ZRDT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: ZRDT 2005
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2007-10-25 (Estimated); Status verified 2007-10

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Rapid Diagnostic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Rapid Diagnostic Test for P. falciparum malaria
  Other Names: Paracheck Pf, Manufactured by Orchid Biomedical Systems, Goa, INDIA.

SUMMARY:
The purpose of this study is to assess performance and cost-effectiveness of rapid diagnostic test(RDT) aided malaria diagnosis versus symptom-based/clinical diagnosis in patients of all ages with reported fever last 48 hours alone in primary health care settings in Zanzibar.

ELIGIBILITY:
Inclusion Criteria:

* Any patient attending the study sites and reporting history of fever within past 48 hours or other symptoms compatible with malaria and giving their informed consent, will be eligible for the study.

Exclusion Criteria:

* Patient's refusal to consent will disqualify participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9346 (Actual)
Dates: Start 2005-02; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Björkman, MD,PhD, Study Director — Karolinska UH; Mwinyi I Msellem, HLSO, Principal Investigator — Karolinska UH
Locations (1):
- Muyuni, Uzini, Kinyasini and Mzambarauni Primary Health Care Units, Zanzibar, Zanzibar, Tanzania

REFERENCES:
- [Derived] Msellem MI, Martensson A, Rotllant G, Bhattarai A, Stromberg J, Kahigwa E, Garcia M, Petzold M, Olumese P, Ali A, Bjorkman A. Influence of rapid malaria diagnostic tests on treatment and health outcome in fever patients, Zanzibar: a crossover validation study. PLoS Med. 2009 Apr 28;6(4):e1000070. doi: 10.1371/journal.pmed.1000070. Epub 2009 Apr 28. PMID 19399156